CLINICAL TRIAL: NCT02772549
Title: Early Diagnosis of Pulmonary Fibrosis
Brief Title: Early Diagnosis of Pulmonary Fibrosis - Diagnostic Delay
Status: Active, not recruiting | Type: Observational
Sponsor: Nils Hoyer (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Nils Hoyer, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: DELAY
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Diagnosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with newly diagnosed IPF are investigated for the diagnostic delay before a diagnosis of IPF is made.

DETAILED DESCRIPTION:
Pulmonary fibrosis can be secondary to connective-tissue disease, environmental exposure, or drug toxicity, but it can also appear sporadically without any known cause, i.e. idiopathic interstitial pneumonitis (IIP). Idiopathic pulmonary fibrosis (IPF) is the commonest IIP and usually follows a rapidly progressive course with a short median survival time.

IPF is often diagnosed after a long diagnostic delay, which also affects the prognosis. As new anti-fibrotic treatments have been approved, and awareness of IPF is rising, the diagnostic delay and its implications can be expected to be changing. Also, the new diagnostic guidelines of 2011 could change the diagnostic delay. In order to reduce the diagnostic delay, it is important to investigate the health care utilization and decisions made by healthcare professionals in the period before the final diagnosis is made.

This study will prospectively include all patients at the two centres in Denmark where patients are treated for IPF and has thus a good opportunity to include the majority of incident cases of IPF in Denmark. Patients are included immediately after the diagnosis which reduces recall bias. The database will include both patient reported data and objective data from national registries and patient records. A main focus is the distribution of the diagnostic delay between patient and different health care providers, and the health care utilization by the patients before a diagnosis of IPF is made. Risk factors for a delayed diagnosis are investigated. The importance of the diagnostic delay for the prognosis and the course of the disease will also be investigated.

The database created in this study will also be used for future research in IPF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF according to international guidelines

Exclusion Criteria:

* Unable to provide written informed consent
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All incident patients with IPF at Gentofte hospital and Aarhus university hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-12 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who fulfil any of the following: disease progression or death | 1 year

SECONDARY OUTCOMES:
Number of patients who fulfill any of the following: decrease in lung function, reduced walking distance at 6 minutes walking test, increased need for supplementary oxygen, hospitalization | 1 year
All-cause and disease-specific mortality | 1 year
Number of respiratory and non-respiratory hospitalizations | 1 year
Decrease in walking distance at the 6 minute walking test | 1 year
Change in St. George Respiratory Questionnaire symptom scores | 1 year
Reduction in diffusion capacity (DLCO) or forced vital capacity (FVC) | 1 year

OTHER OUTCOMES:
Diagnostic delays | 1 year
  Diagnostic delay subdivided into patient related delays and health care related delays.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Hellerup, Copenhagen
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Derived] Hoyer N, Prior TS, Bendstrup E, Wilcke T, Shaker SB. Risk factors for diagnostic delay in idiopathic pulmonary fibrosis. Respir Res. 2019 May 24;20(1):103. doi: 10.1186/s12931-019-1076-0. PMID 31126287